CLINICAL TRIAL: NCT04538898
Title: A Retrospective Study Investigating the Factors Related to Non-tuberculous Mycobacterial Pulmonary Disease in Hong Kong
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Susanna SS Ng, Assistant Professor, Chinese University of Hong Kong
Other Study IDs: NTM in HK_2019
Record Dates: First submitted 2020-08-31; First posted 2020-09-04 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Non-Tuberculous Mycobacterial Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this retrospective study, we aim to investigate the demographic and clinical features of patients with nontuberculous mycobacteria (NTM) lung disease in our hospital and the trends and diversity of NTM species isolated in the period of 2009-2018.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old.
* patients with one or more respiratory isolates (namely, sputum, tracheal aspirates, bronchial washing, bronchial aspirates, bronchial trap and bronchoalveolar lavage) of mycobacteria collected in the Prince of Wales Hospital in the period of 2009-2018.

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Clinical Data Analysis and Reporting System (CDARS) will be queried to identify patients from whom one or more respiratory isolates (namely, sputum, tracheal aspirates, bronchial washing, bronchial aspirates, bronchial trap and bronchoalveolar lavage) of mycobacteria collected in the Prince of Wales Hospital in the period of 2009-2018. Specimen and clinical information is linked through the Clinical Management System (CMS). The clinical history from the CMS will be reviewed to assess the comorbid conditions and baseline demographic information.
  Laboratory reported use of DNA probes for identification of Mycobacterium avium complex (MAC), M. avium, Mycobacterium intracellulare, Mycobacterium kansasii, and Mycobacterium gordonae, high-performance liquid chromatography and biochemical will be used to identify rapid growers. For trend analysis, no changes in methods for species identification during the study periods will be reported.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
diversity of nontuberculous mycobacteria species | 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese University of Hong, Hong Kong, Please Select, Hong Kong

IPD SHARING:
Plan to Share IPD: No